CLINICAL TRIAL: NCT02470923
Title: In-patient Smoking Cessation Intervention Using Counseling, Spirometry and Nicotine Replacement Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Soroka University Medical Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOR-0180-12-CTIL
Record Dates: First submitted 2015-06-10; First posted 2015-06-12 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-05

CONDITIONS: Smoking Cessation
Keywords: Smoking cessation; Nicotine; Spirometry; Internal medicine
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Other): Usual care including medical advice to quit and confrontation with abnormal spirometry results if relevant.
  Interventions: Behavioral: Medical advice
- Group 2 (Other): Intensive counseling (15 minutes) by a smoking cessation counselor including confrontation with abnormal spirometry results if relevant, and follow up for at least 5 weeks after discharge (will be done weekly by phone for five consecutive weeks).
  Interventions: Behavioral: Intensive counseling
- Group 3 (Other): Intensive counseling (15 minutes) by a smoking cessation counselor including confrontation with abnormal spirometry results if relevant, offering and providing nicotine replacement therapy (NRT) and follow up (will be done weekly by phone for five consecutive weeks).
  Interventions: Drug: Nicotine replacement therapy

INTERVENTIONS:
Drug: Nicotine replacement therapy
  Arms: Group 3
Behavioral: Intensive counseling
  Arms: Group 2
Behavioral: Medical advice
  Arms: Group 1

SUMMARY:
The objective of the study is to assess the effect of in-hospital intensive counseling and NRT (nicotine replacement therapy) vs. usual care, on smoking cessation or enrollment to smoking cessation behavioral intervention.

This is prospective randomized clinical trial. The study population will include smokers subjects admitted to internal medicine departments at Soroka University Medical Center.

The study population will be divided randomly into three arms according to intervention intensity (ratio 1:1:1).

DETAILED DESCRIPTION:
Prospective randomized clinical trial. The study population will include smokers subjects admitted to internal medicine departments at Soroka University Medical Center.

The study population will be divided randomly into three arms according to intervention intensity (ratio 1:1:1):

Group 1 - Usual care including medical advice to quit and confrontation with abnormal spirometry results if relevant.

Group 2 - Intensive counseling (15 minutes) by a smoking cessation counselor including confrontation with abnormal spirometry results if relevant, and follow up for at least 5 weeks after discharge (will be done weekly by phone for five consecutive weeks).

Group 3 - Intensive counseling (15 minutes) by a smoking cessation counselor including confrontation with abnormal spirometry results if relevant, offering and providing nicotine replacement therapy (NRT) and follow up (will be done weekly by phone for five consecutive weeks).

All participants will be given a smoking cessation leaflet.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to Internal Medicine at Soroka University Medical Center.
2. Current cigarette smokers (≥ 10 cigarettes per day)
3. Provided written informed consent.

Exclusion Criteria:

1. Substance abuse (except for tobacco).
2. Handicapped or bed ridden patients.
3. Patients who don't speak Hebrew, English, Russian or Arabic.
4. Medically not suitable for NRT-decided by physician on the basis of the patient's medical file.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Composite outcome: •Enrollment to a cessation behavioral intervention program according to participation in first two meetings of group therapy or personal counseling • Smoking cessation validated by CO exhale test<5 ppm | Within six months since discharge
  The need for composite primary outcome based on the hypothesis that in Israel, the best supported way to quit smoking in by participating in group or personal counseling, with 50% success rate of smoking cessation.

CONTACTS AND LOCATIONS:
Locations (1):
- Soroka University Medical Center, Beersheba, Israel

REFERENCES:
- [Result] Rigotti NA, Munafo MR, Stead LF. Smoking cessation interventions for hospitalized smokers: a systematic review. Arch Intern Med. 2008 Oct 13;168(18):1950-60. doi: 10.1001/archinte.168.18.1950. PMID 18852395
- [Result] US Department of Health & Human Services. The Health Consequences of Smoking: A Report of the Surgeon General. 2004. Accessed at www.surgeongeneral.gov/library/smokingconsequences/ on October 31, 2011.
- [Result] Fiore MC, Goplerud E, Schroeder SA. The Joint Commission's new tobacco-cessation measures--will hospitals do the right thing? N Engl J Med. 2012 Mar 29;366(13):1172-4. doi: 10.1056/NEJMp1115176. Epub 2012 Mar 14. No abstract available. PMID 22417200
- [Result] Silagy C, Lancaster T, Stead L, Mant D, Fowler G. Nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2004;(3):CD000146. doi: 10.1002/14651858.CD000146.pub2. PMID 15266423
- [Result] Rigotti NA, Arnsten JH, McKool KM, Wood-Reid KM, Singer DE, Pasternak RC. The use of nicotine-replacement therapy by hospitalized smokers. Am J Prev Med. 1999 Nov;17(4):255-9. doi: 10.1016/s0749-3797(99)00095-1. PMID 10606193
- [Result] McRobbie H, Hajek P. Nicotine replacement therapy in patients with cardiovascular disease: guidelines for health professionals. Addiction. 2001 Nov;96(11):1547-51. doi: 10.1046/j.1360-0443.2001.961115472.x. PMID 11784452
- [Result] Thabane M; COPD Working Group. Smoking cessation for patients with chronic obstructive pulmonary disease (COPD): an evidence-based analysis. Ont Health Technol Assess Ser. 2012;12(4):1-50. Epub 2012 Mar 1. PMID 23074432
- [Result] Kotz D, Wesseling G, Huibers MJ, van Schayck OC. Efficacy of confronting smokers with airflow limitation for smoking cessation. Eur Respir J. 2009 Apr;33(4):754-62. doi: 10.1183/09031936.00116308. Epub 2009 Jan 7. PMID 19129277
- [Result] Stead LF, Lancaster T. Group behaviour therapy programmes for smoking cessation. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD001007. doi: 10.1002/14651858.CD001007.pub2. PMID 15846610
- [Result] Fiore MC, Jaén CR, Baker TB, et al: Clinical practice guideline: treating tobacco use and dependence: 2008 update. Rockville, MD: U.S. Department of Health and Human Services, Public Health Service. Retrieved 2011-02-16.
- [Result] Israel health ministry report 2010, Accessed at: http://www.old.health.gov.il/download/pages/smoke10_290511.pdf